CLINICAL TRIAL: NCT00889902
Title: Molecular Markers in Cervical Cancer Screening in the Feasibility of the Mathematical Markov Model Analysis
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Wuhan University (Other)
Responsible Party: HB Cai, Wuhan University
Other Study IDs: 320.6740
Record Dates: First submitted 2009-04-27; First posted 2009-04-29 (Estimated); Last update posted 2009-04-29 (Estimated); Status verified 2009-04

CONDITIONS: Cervical Cancer
Keywords: Molecular Markers; Cervical Cancer; Screening; Makov
MeSH Terms: conditions — Uterine Cervical Neoplasms

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Cervical exfoliated cells
Oversight: Data Monitoring Committee: Yes

SUMMARY:
The purpose of this study is to:

1. make p16INK4A as a cervical cancer screening of tumor markers, cytology improve existing diagnostic sensitivity, specificity, repeatability and validity, so as to effectively prompted the early discovery and diagnosis of cervical cancer.
2. reduce screening costs, screening and benefits into quantitative evaluation, for our country to develop cervical cancer prevention and control strategy to provide a reliable theoretical basis.

DETAILED DESCRIPTION:
1. To carry out large-scale prospective randomized controlled clinical study to evaluate the "cytological molecular markers Detect + P16INK4A" methods of screening accuracy and reliability, as well as the screening method of the biological effects.
2. Markov set up mathematical model of screening tests to quantify the inputs and the evaluation proceeds. With a view to optimize and perfect a simple, convenient, practical and efficient program of cervical cancer screening.

ELIGIBILITY:
Inclusion Criteria:

* Married women aged 25 to 65-year-old with risk factors
* No tumor and pelvic radiation therapy history
* Non-pregnant women at present

Ages: 25 Years to 65 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: residents of a certain town
Sampling Method: Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2009-04; Primary Completion 2010-06 (Estimated); Study Completion 2011-07 (Estimated)

CONTACTS AND LOCATIONS:
Overall Officials: Hong B Cai, Doctor, Study Director — gynecologic oncology department, Zhongnan Hospital of Wuhan University
Locations (1):
- People'S Hospital, Wufeng County, Hubei, China